CLINICAL TRIAL: NCT05356728
Title: Comparison of the Efficacy of Two Types of Artificial Tears in the Treatment of Dry Eye Disease
Brief Title: Comparison of Two Types of Artificial Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Norwegian Dry Eye Clinic (Other Government)
Collaborators: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyabak vs. Thealoz Duo
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The doctors who examine the patients will not get any information about the choice of artificial tears in each eye.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thealoz Duo (Active Comparator): Thealoz Duo, a combination of trehalose and hyaluronate, will be used on one of the selected eyes of a patient, at least 3 times daily
  Interventions: Drug: Thealoz Duo (combination of trehalose and hyaluronate) eye drop and Hyabak (hyaluronate) eye drop
- Hyabak (Active Comparator): Hyabak, sodium hyaluronate, will be used on the other eye of the patient, at least 3 times daily
  Interventions: Drug: Thealoz Duo (combination of trehalose and hyaluronate) eye drop and Hyabak (hyaluronate) eye drop

INTERVENTIONS:
Drug: Thealoz Duo (combination of trehalose and hyaluronate) eye drop and Hyabak (hyaluronate) eye drop — One of the eyes will be assigned to use Thealoz Duo while the other with Hyabak by using randomisation table

SUMMARY:
Hyaluronic acid (HA), a natural component of the tear film, is a well-established active ingredient in artificial tears and has been reported to improve corneal and conjunctival staining in patients with DED. Thealoz Duo (Laboratoires Thea, Clermont Ferrand, France) is a novel artificial tear preparation containing two active ingredients: trehalose, a naturally occurring disaccharide with anhydrobiotic functions in many organisms, and hyaluronate, a widely distributed anionic glycosaminoglycan polysaccharide with lubricative and water-retaining properties in biological systems. The purpose of the current study is to investigate the effect of the Hyabak and Thealoz Duo in treatment of DED.

DETAILED DESCRIPTION:
The patients will be treated with Thealoz Duo (at least 3 times daily) in one eye and with Hyabak (at least 3 times daily) in the other eye, based on randomization table. Both Hyabak and Thealoz Duo are preservative free. The doctors who examine the patients will not get any information about the choice of artificial tears in each eye. Besides the artificial tears, if necessary, the patients will receive other treatments, for instance, steroids, cyclosporine etc., according to their dry eye severity.

ELIGIBILITY:
Inclusion Criteria:

* Dry Eye Severity Level (DESL) 1-3
* Equivalent between-eye DESL

Exclusion Criteria:

* Ocular infection and/or non-linked inflammation
* Corneal pathology (except KSP)
* Corneal refractive surgery or cataract surgery within 6 months prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Subjective dry eye symptoms | Baseline,
  McMonnies dry eye questionnaire
Subjective dry eye symptoms | 1 month after treatment is initiated
  McMonnies dry eye questionnaire
Subjective dry eye symptoms | 3 months after treatment is initiated
  McMonnies dry eye questionnaire
Subjective dry eye symptoms | Baseline
  Ocular Surface Disease Index (OSDI) dry eye questionnaire
Subjective dry eye symptoms | 1 month after treatment is initiated
  Ocular Surface Disease Index (OSDI) dry eye questionnaire
Subjective dry eye symptoms | 3 months after treatment is initiated
  Ocular Surface Disease Index (OSDI) dry eye questionnaire

SECONDARY OUTCOMES:
Fluorescein tear film break up time | Baseline
  Unit: seconds
Fluorescein tear film break up time | 1 month after treatment is initiated
  Unit: seconds
Fluorescein tear film break up time | 3 months after treatment is initiated
  Unit: seconds
Schirmer test | Baseline
  Without anaesthesia, recorded as mm in length of wetting after 5min
Schirmer test | 1 month after treatment is initiated
  Without anaesthesia, recorded as mm in length of wetting after 5min
Schirmer test | 3 months after treatment is initiated
  Without anaesthesia, recorded as mm in length of wetting after 5min
Ocular surface staining | Baseline
  Fluorescein staining at the conjunctiva and cornea. Recorded using oxford scheme, range 0-15
Ocular surface staining | 1 month after treatment is initiated
  Fluorescein staining at the conjunctiva and cornea. Recorded using oxford scheme, range 0-15
Ocular surface staining | 3 months after treatment is initiated
  Fluorescein staining at the conjunctiva and cornea. Recorded using oxford scheme, range 0-15
Tear film osmolarity | Baseline
  Unit: Osm/L
Tear film osmolarity | 1 month after treatment is initiated
  Unit: Osm/L
Tear film osmolarity | 3 month after treatment is initiated
  Unit: Osm/L
Meibum expressibility | Baseline
  Evaluated by application of light pressure using cotton tips on the central five MGs of the lower eyelid. Expression was graded according to the number of the MGs with meibum secretion under pressure: grade 0: 5 glands; grade 1: 3-4 glands; grade 2: 1-2 glands; grade 3: 0 gland
Meibum expressibility | 1 month after treatment is initiated
  Evaluated by application of light pressure using cotton tips on the central five MGs of the lower eyelid. Expression was graded according to the number of the MGs with meibum secretion under pressure: grade 0: 5 glands; grade 1: 3-4 glands; grade 2: 1-2 glands; grade 3: 0 gland
Meibomian gland functionality | 3 months after treatment is initiated
  Meibum expressibility and quality
Meibum quality | Baseline
  The quality of the meibum that was secreted from each gland was graded as following: 0, clear; 1, cloudy; 2, cloudy with particles; and 3, toothpaste like. The sum of the score of the central 8 glands in the lower eyelid will be recorded
Meibum quality | 1 month after treatment is initiated
  The quality of the meibum that was secreted from each gland was graded as following: 0, clear; 1, cloudy; 2, cloudy with particles; and 3, toothpaste like. The sum of the score of the central 8 glands in the lower eyelid will be recorded
Meibum quality | 3 months after treatment is initiated
  The quality of the meibum that was secreted from each gland was graded as following: 0, clear; 1, cloudy; 2, cloudy with particles; and 3, toothpaste like. The sum of the score of the central 8 glands in the lower eyelid will be recorded
Patient´s subjective evaluation of preference | 1 month after the treatment is initiated
  Patients will be asked about which artificial tear they prefer
Patient´s subjective evaluation of preference | 3 months after the treatment is initiated
  Patients will be asked about which artificial tear they prefer
Luminex | Baseline
  A multiplex Luminex® bead-based assay will be used to analyze cytokines from the tear samples. The cytokines to be analysed include 27 different cytokines, including interleukin 1b (IL-1b), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17A, IL-1 receptor antagonist (IL-1ra), eotaxin, basic fibroblast growth factor (bFGF/FGF2), granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFN-γ), interferon gamma-induced protein 10 (IP-10), monocyte chemoattractant protein 1 (MCP-1), macrophage inflammatory protein 1α (MIP-1α/CCL3), MIP-1b, platelet-derived growth factor bb (PDGF-BB), regulated-on-activation normal T cell expressed and secreted (Rantes), tumor necrosis factor alpha (TNF-α), and vascular endothelial growth factor (VEGF).
Luminex | 1 month after treatment is initiated
  A multiplex Luminex® bead-based assay will be used to analyze cytokines from the tear samples. The cytokines to be analysed include 27 different cytokines, including interleukin 1b (IL-1b), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17A, IL-1 receptor antagonist (IL-1ra), eotaxin, basic fibroblast growth factor (bFGF/FGF2), granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFN-γ), interferon gamma-induced protein 10 (IP-10), monocyte chemoattractant protein 1 (MCP-1), macrophage inflammatory protein 1α (MIP-1α/CCL3), MIP-1b, platelet-derived growth factor bb (PDGF-BB), regulated-on-activation normal T cell expressed and secreted (Rantes), tumor necrosis factor alpha (TNF-α), and vascular endothelial growth factor (VEGF).
Luminex | 3 months after treatment is initiated
  A multiplex Luminex® bead-based assay will be used to analyze cytokines from the tear samples. The cytokines to be analysed include 27 different cytokines, including interleukin 1b (IL-1b), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17A, IL-1 receptor antagonist (IL-1ra), eotaxin, basic fibroblast growth factor (bFGF/FGF2), granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFN-γ), interferon gamma-induced protein 10 (IP-10), monocyte chemoattractant protein 1 (MCP-1), macrophage inflammatory protein 1α (MIP-1α/CCL3), MIP-1b, platelet-derived growth factor bb (PDGF-BB), regulated-on-activation normal T cell expressed and secreted (Rantes), tumor necrosis factor alpha (TNF-α), and vascular endothelial growth factor (VEGF).

CONTACTS AND LOCATIONS:
Locations (1):
- The Norwegian Dry Eye Clinic, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No